CLINICAL TRIAL: NCT03398525
Title: Effect of a Musical Intervention in the Intensive Care Unit During the Implantation of a Central Venous Access or a Dialysis Catheter: A Prospective, Randomized Pilot Study
Brief Title: Musical Intervention and Patient's Anxiety During Central Venous Catheter Insertion in the Intensive Care Unit
Acronym: MUSIC-CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHRO-2017-11; IDRCB number: 2017-A02536-47 (Other: French Government)
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Anxiety; Pain
Keywords: central venous catheter; intensive care; music therapy
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: randomization with 1:1 allocation ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): After patient information, appropriate skin antisepsis according to local procedures, surgical hand antisepsis by the operator, use of sterile drapes, gowns and gloves, insertion of a central venous catheter after after local anesthesia with 2% lidocaine, using ultrasound guidance.
  Interventions: Other: usual care
- Musical intervention (Experimental): After patient information, appropriate skin antisepsis according to local procedures, surgical hand antisepsis by the operator, use of sterile drapes, gowns and gloves, insertion of a central venous catheter after after local anesthesia with 2% lidocaine, using ultrasound guidance.
  In addition, a U-shaped music program (MUSIC CARE, trade mark) will be delivered to the patient through headphones throughout the catheter insertion procedure beginning with the operator's hand washing and ending once the dressing is put on the catheter insertion site.
  Interventions: Other: usual care; Other: Musical intervention

INTERVENTIONS:
Other: usual care — usual care following local standard operational procedures
Other: Musical intervention — Musical intervention using a marketed music program validated for music therapy
  Arms: Musical intervention

SUMMARY:
Intensive care unit patients who have to undergo central venous catheter insertion and are able to hear explanations and to gave consent, will be randomized to either usual care during catheter insertion or to a musical intervention added to usual care.

The primary objective will be to assess the patient's anxiety just after catheter insertion. Secondary outcome measures will be the patient-reported pain, the duration of catheter insertion, and the need for additional anxiolytic or sedative drugs during catheter insertion.

DETAILED DESCRIPTION:
Patient informed consent will be obtained before any other study specific procedure.

Computer-generated randomization with 1:1 allocation ratio will be stratified by the site of catheter insertion (superior vena cava or femoral), and by the ventilatory status (patient mechanically ventilated or not). Block size, not known by the investigators, of 4 or 6 will be used. Randomization group for each patient will be kept concealed into sealed opaque envelops until inclusion once consent obtained.

Anxiety, the primary outcome measure, and pain related to the catheter insertion will be assessed using two distinct Visual Analogic Scales.

In the usual care group, the catheter will be inserted using the Seldinger method, under local anesthesia with 2% lidocaine, with ultrasound guidance, after proper skin antisepsis, surgical operator's hand washing and antisepsis, and use of sterile drapes, gowns and gloves.

In the intervention group, in addition to the usual care procedures as described above, a musical U-shaped session will be delivered to the patient through headphones, using a tablet computer and the "MUSIC CARE" music program, a validated program for use in health care.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized in the intensive care unit or high-dependency unit
* patient for whom a central venous catheter insertion is envisaged
* patient capable of hearing and understanding explanations and able to consent

Exclusion Criteria:

* severe hearing loss
* allergy to local anesthetic drug
* pregnancy
* lack of social security number
* patient under guardianship
* previous participation to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
anxiety assessed using a visual analog scale (VAS) | 30 minutes
  self-reported patient's anxiety assessed using a 100mm-visual analog scale, extending from 0 mm ("no anxiety") to 100 mm ("worst anxiety ever experienced")

SECONDARY OUTCOMES:
pain assessed using a visual analog scale (VAS) | 30 minutes
  self-reported patient's pain assessed using a 100mm-visual analog scale, extending from 0 mm ("no pain") to 100 mm ("the worst pain possible")
duration of the catheter insertion | 10-30 min
  started with local anesthesia and ending with the application of the dressing on catheter insertion site.

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Ahn Nay, MD, Principal Investigator — CHR Orléans, France
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacquier S, Nay MA, Muller G, Muller L, Mathonnet A, Lefevre-Benzekri D, Bretagnol A, Barbier F, Kamel T, Runge I, Skarzynski M, Sauvage B, Boulain T. Effect of a Musical Intervention During the Implantation of a Central Venous Catheter or a Dialysis Catheter in the Intensive Care Unit: A Prospective Randomized Pilot Study. Anesth Analg. 2022 Apr 1;134(4):781-790. doi: 10.1213/ANE.0000000000005696. PMID 35299213